CLINICAL TRIAL: NCT05512572
Title: Therapeutic Efficacy of Intense Pulsed Light in the Treatment of Chalazion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0563
Record Dates: First submitted 2022-08-21; First posted 2022-08-23 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2021-09

CONDITIONS: Chalazion
MeSH Terms: conditions — Chalazion | interventions — Conservative Treatment; Curettage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Receiving IPL-MGD treatment.
  Interventions: Device: IPL
- Control group (Active Comparator): Another set of age, sex and diagnosis matched consecutive cases of chalazion, who received conservative treatment or excision with curettage but without IPL-MGX treatment as a control (Non-IPL group).
  Interventions: Procedure: Conservative treatment or excision with curettage

INTERVENTIONS:
Device: IPL — intense pulsed light
  Arms: Experimental group
Procedure: Conservative treatment or excision with curettage — conservative treatment or excision with curettage but without IPL-MGX treatment as a control
  Arms: Control group

SUMMARY:
Study method: This test screened the subjects first, and proposed to include 50 subjects with primary or recurrent eyelid plate gland cysts without obvious surgical indications. All subjects underwent three strong pulsed light therapy combined with eyelid plate gland massage, treatment of local anesthesia eye drops, and metal pads were placed in conjunctival sac protection. Eye protection, using the M22 strong pulsed light small optical treatment head of the medical company, energy selection 14-16J/cm2, laser position is selected on the upper and lower eyelids, 3mm away from the root of the eyelashes. Each interval is 3 weeks. Eye-related examinations were performed before treatment and 3 times after treatment. The evaluation content included: ocular surface, slit lamp observation, anterior segment photography, intraocular pressure, vision, corneal fluorescein staining, tear film rupture time, eyelid plate gland evaluation, eyelid plate gland cyst relief, eyelid plate gland cyst recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients had primary or recurrent eyelid plate gland cyst without obvious surgical indications

Exclusion Criteria:

* (1) any intraocular inflammation, ocular infection, allergy, ocular surgery, or ocular trauma in the past 6 months; (2) any eyelid diseases or structural abnormality; (3) any systematic diseases may lead to dry eye or MGD; (4) skin cancer or pigmented lesion in the treatment zone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2023-08-23 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of chalazia | An average of 1 year
  The recurrence of the chalazia

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University Hospital, Hangzhou, Zhejiang, China